CLINICAL TRIAL: NCT04912804
Title: Perceived Health After Hospitalization for COVID-19
Acronym: PRO-COVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DEVILLIERS AOIc 2020
Record Dates: First submitted 2021-06-02; First posted 2021-06-03 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: COVID-19, Post-hospitalization, Disease Impact
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Patient: Patient discharged from a conventional short-stay hospitalization unit.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — SF-12, GHQ-12 and HAQ

SUMMARY:
There are currently no precise data available on the impact of COVID-19 on the daily life of patients after hospitalization. For the moment, studies have only demonstrated a strong impact of the diagnosis on the domains of quality of life explored by the MOS-SF36 questionnaire and the PHQ-9 depression score. Concerning the impact of COVID-19 disease after conventional hospitalization, field reports indicate extremely intense fatigue and a major physical impact lasting several weeks

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient with a diagnosis of COVID-19 confirmed by PCR and/or CT scan
* Patient hospitalized in a short stay unit (excluding intensive care and rehabilitation) for a COVID-19 infection
* Patient providing oral consent to participate in the study
* Patient able to understand and answer the questionnaires used
* Patient able to answer the questions on an electronic device and to receive requests by email and/or SMS
* Patient who has electronic equipment at home and an Internet subscription allowing him/her to answer the questionnaires online

Exclusion Criteria:

* Patient under guardianship, curatorship or a measure of judicial safeguard

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with COVID-19 discharged from a conventional short-stay hospital ward.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-05-22 (Actual); Study Completion 2021-05-22 (Actual)

PRIMARY OUTCOMES:
Time to PASS and CID in patients discharged from conventional hospitalization for COVID-19 disease | Through study completion, an average of 6 months
The value of perceived health scores in patients who achieved PASS and MCII | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France